CLINICAL TRIAL: NCT02171806
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Inhalative Doses (2.5 μg, 10 μg, and 30 μg) of BI 1744 CL for 14 Days in Healthy Male and Female Volunteers (Doubleblind, Randomised, Placebo Controlled [at Each Dose Level] Study)
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of BI 1744 CL in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1222.2
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — olodaterol

ARMS (3):
- BI 1744 CL multiple rising doses (Experimental)
  Interventions: Drug: BI 1744 CL
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BI 1744 CL medium dose, females (Experimental)
  Interventions: Drug: BI 1744 CL

INTERVENTIONS:
Drug: BI 1744 CL
  Arms: BI 1744 CL medium dose, females; BI 1744 CL multiple rising doses
Drug: Placebo
  Arms: Placebo

SUMMARY:
To investigate safety, tolerability, pharmacokinetics and pharmacodynamics of BI 1744 CL

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female based upon a complete medical history, including the physical examination, regarding vital signs (blood pressure (BP), pulse rate (PR)), 12-lead ECG measurement, and clinical laboratory tests. There is no finding deviating from normal and of clinical relevance. There is no evidence of a clinically relevant concomitant disease.
* Age ≥21 and ≤50 years
* BMI ≥18.5 and <30 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR, and ECG measurements) deviating from normal and of clinical relevance
* Evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to the drug or its excipients) as judged clinically relevant by the investigator
* Intake of drugs with a long half-life (>24 hours) within at least 1 month or less than 10 half-lives of the respective drug prior to randomisation
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to randomisation
* Participation in another trial with an investigational drug within 2 months prior to randomisation
* Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking on trial days as judged by the investigator
* Alcohol abuse (more than 60 g alcohol a day)
* Drug abuse
* Blood donation (more than 100 mL blood within 4 weeks prior to randomisation or during the trial)
* Excessive physical activities within 1 week prior to randomisation or during the trial
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of the study centre

The following exclusion criteria are specific for this study due to the known class side effect profile of ß2-mimetics:

* Asthma or history of pulmonary hyperreactivity
* Hyperthyrosis
* Allergic rhinitis in need of treatment
* Clinically relevant cardiac arrhythmia
* Paroxysmal tachycardia (>100 beats per minute).

For female subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception e.g. oral contraception, sterilisation, IUD (intrauterine device). Females who are not surgically sterile will be asked to additionally use barrier contraception methods (e.g. condoms) prior to administration of study medication, during the study and at least 2 months after release from the study.
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2006-01; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with clinically significant changes in physical examination | Baseline, day 32 (end-of-study examination)
Number of patients with clinically significant changes in vital signs | Baseline, up to day 32
Number of patients with clinically significant changes in 12-lead ECG (Electrocardiogram) | Baseline, up to day 32
Number of patients with abnormal changes in laboratory tests | Baseline, up to day 32
Changes in airway resistance (Raw) measured by body plethysmography | Baseline, up to day 32
Changes in tremormetry parameters | Baseline, up to day 32
Number of patients with adverse events | Up to day 32
Assessment of tolerability by the investigator on a 4-point scale | Day 32 (end-of-study examination)

SECONDARY OUTCOMES:
Cmax (maximum concentration of the analyte in plasma) | Up to 408 hours after drug administration
tmax (time from dosing to maximum concentration) | Up to 408 hours after drug administration
AUC (area under the concentration-time curve of the analyte in plasma at different time points) | Up to 408 hours after drug administration
Aet1-t2(amount of analyte that is eliminated in urine from the time point t1 to time point t2) | Up to 384 hours after drug administration
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | Up to 384 hours after drug administration
%AUCtz-∞ (the percentage of the AUC 0-∞ that is obtained by extrapolation) | Up to 408 hours after drug administration
λz (terminal rate constant of the analyte in plasma) | Up to 408 hours after drug administration
t½ (terminal half-life of the analyte in plasma) | Up to 408 hours after drug administration
MRTih (mean residence time of the analyte in the body after inhalation) | Up to 408 hours after drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | Up to 408 hours after drug administration
Vz/F (apparent volume of distribution of the analyte during the terminal phase λz following an extravascular dose) | Up to 408 hours after drug administration
CLR,t1-t2 (renal clearance of the analyte in plasma from the time point t1 until the time point t2) | Up to 408 hours after drug administration
RA,Cmax,14 based on Cmax (Accumulation ratio of the analyte in plasma after multiple dose administration over a uniform dosing interval τ) | Up to 408 hours after drug administration
RA,AUC,14 based on AUC0-τ | Up to 408 hours after drug administration
Cmin,ss (minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | Up to 408 hours after drug administration
Cpre,ss (predose concentration of the analyte in plasma at steady state immediately before administration of the next dose) | Up to 408 hours after drug administration
Linearity Index (LI) | Up to 408 hours after drug administration